CLINICAL TRIAL: NCT02301988
Title: A Phase II Randomized, Double-Blind, Study of Ipatasertib (GDC-0068), an Inhibitor to AKT, in Combination With Paclitaxel as Neoadjuvant Treatment for Patients With Early Stage Triple Negative Breast Cancer
Brief Title: A Study of Ipatasertib (GDC-0068) in Combination With Paclitaxel as Neoadjuvant Treatment for Participants With Early Stage Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: SOLTI Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO29505; 2014-003029-16 (EudraCT Number)
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Results first posted 2018-09-20 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ipatasertib; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ipatasertib + Paclitaxel (Experimental): Participants will receive ipatasertib orally daily on Days 1-21 of each 28-day cycle for 3 cycles and paclitaxel intravenous (IV) infusion every week (QW) for 3 cycles (12 total doses).
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel
- Placebo + Paclitaxel (Placebo Comparator): Participants will receive placebo (matching to ipatasertib) orally daily on Days 1-21 of each 28-day cycle for 3 cycles and paclitaxel IV infusion QW for 3 cycles (12 total doses).
  Interventions: Drug: Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: Ipatasertib — Ipatasertib will be administered at a dose of 400 milligrams (mg) orally daily on Days 1-21 of each 28-day cycle for 3 cycles.
  Other Names: GDC-0068
  Arms: Ipatasertib + Paclitaxel
Drug: Paclitaxel — Paclitaxel will be administered at a dose of 80 milligrams per square meter (mg/m^2) as IV infusion QW for 3 cycles.
Drug: Placebo — Participants will receive placebo (matching to ipatasertib) orally daily on Days 1-21 of each 28-day cycle for 3 cycles.
  Arms: Placebo + Paclitaxel

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter, pre-operative Phase II study designed to estimate the efficacy of ipatasertib combined with paclitaxel chemotherapy versus placebo combined with paclitaxel chemotherapy in women with Stage Ia - IIIa triple-negative breast adenocarcinoma. The anticipated time on study treatment is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal or postmenopausal women
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically documented, Stage Ia to operable Stage IIIa, triple-negative carcinoma of the breast with primary tumor greter than or equal to (>/=) 1.5 centimeters (cm) in largest diameter (cT1-3) by MRI
* Adequate hematologic and organ function within 14 days before the first study treatment
* Availability of tumor tissue from formalin-fixed, paraffin-embedded (FFPE) core biopsy of breast primary tumor
* For female participants of childbearing potential, agreement to use highly effective form(s) of contraception for the duration of the study and for at least 6 months after last dose of study treatment

Exclusion Criteria:

* Known human epidermal growth factor 2 (HER2)-positive, estrogen receptor (ER)-positive, or progesterone receptor (PgR)-positive breast cancer
* Any prior treatment for the current primary invasive breast cancer
* Participants with cT4 or cN3 stage breast tumors
* Metastatic (Stage IV) breast cancer
* Bilateral invasive breast cancer
* Multicentric breast cancer
* Any disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the participant at high risk from treatment complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (42):
- United States (16):
  - Arizona Oncology Associates, PC-CASA, Tucson, Arizona
  - Sansum Medical Clinic, Inc., Santa Barbara, California
  - Rocky Mountain Cancer Center - Lakewood (West), Lakewood, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mass General/North Shore Cancer, Danvers, Massachusetts
  - Nebraska Cancer Specialists; Oncology Hematology West, PC, Omaha, Nebraska
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Northwest Cancer Specialists - Portland (NE Hoyt St), Portland, Oregon
  - Roper Bon Secours St. Francis Cancer Center, Charleston, South Carolina
  - Texas Oncology, Austin, Texas
  - Texas Oncology Cancer Center, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Houston (Gessner), Houston, Texas
  - Texas Oncology-Tyler, Irving, Texas
  - South Texas Cancer Center - McAllen, McAllen, Texas
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
- Portugal (3):
  - IPO de Lisboa; Servico de Oncologia Medica, Lisbon
  - Hospital Beatriz Angelo; Departamento de Oncologia, Loures
  - IPO do Porto; Servico de Oncologia Medica, Porto
- Spain (23):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Son Llatzer; Servicio de Oncologia, Palma de Mallorca, Balearic Islands
  - Hospital Provincial de Castellon; Servicio de Oncologia, Castellon, Castellon
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Oncologia, Santiago de Compostela, LA Coruña
  - Hospital Universitari de Lleida Arnau de Vilanova, Lleida, Lerida
  - Hospital Universitario Fundación Alcorcón, Alcorcón (Madrid), Madrid
  - Hospital Rey Juan Carlos; Pharmacy, Móstoles, Madrid
  - Hospital Regional Universitario Carlos Haya; hospital Materno Infantil, servicio de Farmacia, Málaga, Malaga
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital Universitari Sant Joan de Reus; Servicio de Oncologia, Reus, Tarragona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital San Pedro De Alcantara; Servicio de Oncologia, Cáceres
  - Hospital Universitari de Girona Dr. Josep Trueta; Servicio de Oncologia, Girona
  - Centro Oncologico MD Anderson International Espana, Madrid
  - Fundacion Jimenez Diaz; Servicio de Oncologia, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Centro Integral Oncologico Clara Campal (CIOCC); Dirección Médica, Madrid
  - Hospital Quiron de Madrid; Servicio de Oncologia, Madrid
  - Hospital Universitario de Fuenlabrada; Servicio de Oncologia, Madrid
  - Hospital Virgen del Rocio, Seville
  - Hospital Clinico Universitario; Oncologia, Valencia

REFERENCES:
- [Derived] Oliveira M, Saura C, Nuciforo P, Calvo I, Andersen J, Passos-Coelho JL, Gil Gil M, Bermejo B, Patt DA, Ciruelos E, de la Pena L, Xu N, Wongchenko M, Shi Z, Singel SM, Isakoff SJ. FAIRLANE, a double-blind placebo-controlled randomized phase II trial of neoadjuvant ipatasertib plus paclitaxel for early triple-negative breast cancer. Ann Oncol. 2019 Aug 1;30(8):1289-1297. doi: 10.1093/annonc/mdz177. PMID 31147675

RESULTS

PARTICIPANT FLOW:
Groups:
- Ipatasertib + Paclitaxel: Participants received ipatasertib orally daily on Days 1-21 of each 28-day cycle for 3 cycles and paclitaxel intravenous (IV) infusion every week (QW) for 3 cycles (12 total doses).
- Placebo + Paclitaxel: Participants received placebo (matching to ipatasertib) orally daily on Days 1-21 of each 28-day cycle for 3 cycles and paclitaxel IV infusion QW for 3 cycles (12 total doses).
Period: Overall Study
Arm/Group | Ipatasertib + Paclitaxel | Placebo + Paclitaxel
Started | 76 | 75
Completed | 66 | 66
Not Completed | 10 | 9
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 2 | 2
Not completed — Unknown Reason | 1 | 3
Not completed — Lack of Efficacy | 3 | 2
Not completed — Death | 1 | 0
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all randomized participants, with participants allocated to the treatment arms to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipatasertib + Paclitaxel | Placebo + Paclitaxel | Total
Number analyzed (Participants) | 76 | 75 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (10.9) | 53.8 (12.0) | 53.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 75 | 151
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 3 | 5
  White | 71 | 70 | 141
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pathological Complete Response (pCR) in Breast and Axilla as Defined by ypT0/Tis ypN0 in the American Joint Committee on Cancer Staging System (in All Participants)
Description: pCR was defined by ypT0/Tis ypN0 in the American Joint Committee on Cancer (AJCC) Staging System with the following determination for breast and axilla by local pathology laboratory evaluation: T0: no evidence of primary tumor; Tis: early cancer that has not spread to neighboring tissue and N0: no cancer found in the lymph nodes.
Time Frame: Surgery visit (at approximately Weeks 14 to 19)
Population: The ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipatasertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 76 | 75
percentage of participants | 17.1 [9.82 to 27.25] | 13.3 [6.58 to 22.86]
Statistical Analysis 1: Comparison: Ipatasertib + Paclitaxel vs Placebo + Paclitaxel; Unstratified Analysis; Test type: Superiority; p = 0.519, Chi-squared; Difference in Response Rates = 3.77, 95% CI [-8.99 to 16.54] — 95% CI for difference in rates were constructed using normal approximation (Wald) with continuity correction

2. Primary Outcome: Percentage of Participants With pCR in Breast and Axilla as Defined by ypT0/Tis ypN0 in the American Joint Committee on Cancer Staging System (in Participants Who Have Phosphatase and Tensin Homolog [PTEN]-Low Tumors)
Description: pCR was defined by ypT0/Tis ypN0 in the AJCC Staging System with the following determination for breast and axilla by local pathology laboratory evaluation: T0: no evidence of primary tumor; Tis: early cancer that has not spread to neighboring tissue and N0: no cancer found in the lymph nodes.
Time Frame: Surgery visit (at approximately Weeks 14 to 19)
Population: The ITT population included all randomized participants who have PTEN-low tumors.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipatasertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 19 | 16
percentage of participants | 15.8 [4.45 to 38.36] | 12.5 [2.27 to 35.43]
Statistical Analysis 1: Comparison: Ipatasertib + Paclitaxel vs Placebo + Paclitaxel; Unstratified analysis; Test type: Superiority; p = 0.7817, Chi-squared; Difference in response rates = 3.29, 95% CI 2-sided [-25.52 to 32.10] — 95% CI for difference in rates were constructed using normal approximation (Wald) with continuity correction

3. Secondary Outcome: Percentage of Participants With pCR in Breast as Defined by ypT0/Tis in the American Joint Committee on Cancer Staging System (in All Participants)
Description: pCR was defined by ypT0/Tis in the AJCC Staging System with the following determination for breast by local pathology laboratory evaluation: T0: no evidence of primary tumor; Tis: early cancer that has not spread to neighboring tissue.
Time Frame: Surgery visit (at approximately Weeks 14 to 19)
Population: The ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipatasertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 76 | 75
percentage of participants | 22.4 [14.33 to 33.31] | 14.7 [7.98 to 24.04]
Statistical Analysis 1: Comparison: Ipatasertib + Paclitaxel vs Placebo + Paclitaxel; Unstratified analysis; Test type: Superiority; p = 0.2234, Chi-squared; Difference in Response Rates = 7.70, 95% CI 2-sided [-5.95 to 21.35] — 95% CI for difference in rates were constructed using normal approximation (Wald) with continuity correction

4. Secondary Outcome: Percentage of Participants With pCR in Breast as Defined by ypT0/Tis in the American Joint Committee on Cancer Staging System (in Participants Who Have PTEN-low Tumors)
Description: as for outcome 3
Time Frame: Surgery visit (at approximately Weeks 14 to 19)
Population: The ITT population included all randomized participants who have PTEN-low tumors.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipatasertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 19 | 16
percentage of participants | 15.8 [4.45 to 38.36] | 18.8 [5.31 to 42.94]
Statistical Analysis 1: Comparison: Ipatasertib + Paclitaxel vs Placebo + Paclitaxel; Unstratified analysis; Test type: Superiority; p = 0.8169, Chi-squared; Difference in response rates = -2.96, 95% CI 2-sided [-33.91 to 27.99] — 95% CI for difference in rates were constructed using normal approximation (Wald) with continuity correction

5. Secondary Outcome: Percentage of Participants With Objective Tumor Response by Magnetic Resonance Imaging (MRI), As Assessed by Investigator Per the Modified Response Evaluation Criteria in Solid Tumors (RECIST) (in All Participants)
Description: Objective tumor response (OR) was based on criteria related to changes in size of target lesions according to modified RECIST. Target lesions were selected on the basis of their size (lesions with the longest diameter) as well as the feasibility of reproducible repeated measurements. OR was the sum of complete response (CR) and partial response (PR). CR: disappearance of all target lesions. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Screening up to disease progression or death (assessed at screening, pre-surgical visit [approximately Weeks 10-12], early termination visit [up to Week 16])
Population: The ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipatasertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 76 | 75
percentage of participants | 67.1 [55.86 to 77.46] | 56.0 [44.46 to 66.84]
Statistical Analysis 1: Comparison: Ipatasertib + Paclitaxel vs Placebo + Paclitaxel; Unstratified analysis; Test type: Superiority; p = 0.1607, Chi-squared; Difference in response rate = 11.11, 95% CI [-5.64 to 27.85] — 95% CI for difference in rates were constructed using normal approximation (Wald) with continuity correction

6. Secondary Outcome: Percentage of Participants With Objective Tumor Response by MRI, As Assessed by Investigator Per Modified RECIST (in Participants Who Have PTEN-low Tumors)
Description: ORR was based on criteria related to changes in size of target lesions according to modified RECIST. Target lesions were selected on the basis of their size (lesions with the longest diameter) as well as the feasibility of reproducible repeated measurements. ORR was the sum of complete response (CR) and partial response (PR). CR: disappearance of all target lesions. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 5
Population: The ITT population included all randomized participants who have PTEN-low tumors.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipatasertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 19 | 16
percentage of participants | 73.7 [50.00 to 89.01] | 50.0 [27.20 to 72.80]
Statistical Analysis 1: Comparison: Ipatasertib + Paclitaxel vs Placebo + Paclitaxel; Unstratified Analysis; Test type: Superiority; p = 0.1486, Chi-squared; Difference in Response Rates = 23.68, 95% CI 2-sided [-13.57 to 60.94] — 95% CI for difference in rates were constructed using normal approximation (Wald) with continuity correction

7. Secondary Outcome: Percentage of Participants With pCR in Breast and Axilla as Defined by ypT0/Tis ypN0 in the American Joint Committee on Cancer Staging System (in Participants Who Are Akt Diagnostic Positive [Dx+])
Description: as for outcome 2
Time Frame: Surgery visit (at approximately Weeks 14 to 19)
Population: The ITT population included all randomized participants who are Akt Dx+.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipatasertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 28 | 34
percentage of participants | 17.9 [7.31 to 35.71] | 11.8 [4.12 to 27.19]
Statistical Analysis 1: Comparison: Ipatasertib + Paclitaxel vs Placebo + Paclitaxel; Test type: Superiority; p = 0.4980, Chi-squared; Difference in Response Rates = 6.09, 95% CI 2-sided [-15.01 to 27.20] — 95% CI for difference in rates were constructed using normal approximation (Wald) with continuity correction method

8. Secondary Outcome: Percentage of Participants With pCR in Breast as Defined by ypT0/Tis in the American Joint Committee on Cancer Staging System (in Participants Who Are Akt Dx+)
Description: as for outcome 3
Time Frame: Surgery visit (at approximately Weeks 14 to 19)
Population: The ITT population included all randomized participants who are Akt Dx+.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipatasertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 28 | 34
percentage of participants | 21.4 [9.77 to 40.58] | 11.8 [4.12 to 27.19]
Statistical Analysis 1: Comparison: Ipatasertib + Paclitaxel vs Placebo + Paclitaxel; Test type: Superiority; p = 0.3032, Chi-squared; Difference in Response Rates = 9.66, 95% CI [-12.25 to 31.58] — 95% CI for difference in rates were constructed using normal approximation (Wald) with continuity correction method

9. Secondary Outcome: Percentage of Participants With pCR According to American Joint Committee on Cancer Staging System, by Breast Cancer Subtype
Description: pCR was defined by ypT0/Tis in the AJCC Staging System with the following determination for breast subtypes by local pathology laboratory evaluation: T0: no evidence of primary tumor; Tis: early cancer that has not spread to neighboring tissue. The intrinsic molecular subtypes of breast cancer included here are luminal A (LumA), Her-2, basal-like, normal and unknown.
Time Frame: Surgery visit (at approximately Weeks 14 to 19)
Population: The ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ipatasertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 76 | 75
percentage of participants
  Unknown: number analyzed (Participants) | 27 | 32
  Unknown | 18.5 | 21.9
  Basal: number analyzed (Participants) | 41 | 37
  Basal | 22.0 | 10.8
  Her2: number analyzed (Participants) | 6 | 3
  Her2 | 33.3 | 0
  LumA: number analyzed (Participants) | 0 | 1
  LumA |  | 0
  Normal: number analyzed (Participants) | 2 | 2
  Normal | 50.0 | 0

10. Secondary Outcome: Percentage of Participants With Response to Undergoing Breast Conserving Surgery (BCS) Among Participants With T2 or T3 Tumors
Description: After neoadjuvant treatment, the number of patients who is appropriate for breast conserving surgery is reported as a measure of efficacy of the treatment to shrink the tumor enough for patients to benefit from less aggressive surgical management. Breast-conserving surgery was defined as removal of part of the breast tissue during surgery. T2 or T3 in the AJCC Staging System were defined as follows: T2: tumor was more than 2 centimeter (cm) but no more than 5 cm across; T3: tumor was larger than 5 cm across.
Time Frame: Surgery visit (at approximately Weeks 14 to 19)
Population: The ITT population included all randomized participants with T2 or T3 Tumors.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipatasertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 62 | 63
percentage of participants | 64.5 [51.93 to 76.26] | 60.3 [47.20 to 71.74]
Statistical Analysis 1: Comparison: Ipatasertib + Paclitaxel vs Placebo + Paclitaxel; Test type: Superiority; p = 0.6280, Chi-squared; Difference in Response Rates = 4.20, 95% CI 2-sided [-14.37 to 22.76] — 95% CI for difference in rates were constructed using normal approximation (Wald) with continuity correction method

11. Secondary Outcome: Percentage of Participants With Response to Conversion to BCS Among Participants With T2 or T3 Tumors
Description: as for outcome 10
Time Frame: From screening to surgery visit (at approximately Weeks 14 to 19)
Population: The ITT population included all randomized participants with T2 or T3 Tumors with response to conversion to BCS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipatasertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 12 | 16
percentage of participants | 33.3 [12.29 to 65.11] | 25 [9.03 to 50.00]
Statistical Analysis 1: Comparison: Ipatasertib + Paclitaxel vs Placebo + Paclitaxel; Test type: Superiority; p = 0.6291, Chi-squared; Difference in Response Rates = 8.33, 95% CI 2-sided [-33.04 to 49.71] — 95% CI for difference in rates were constructed using normal approximation (Wald) with continuity correction method

12. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Screening up to Week 24
Population: The safety population was identical to the ITT population and included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ipatasertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 76 | 75
percentage of participants | 100 | 98.7

13. Secondary Outcome: Plasma Concentrations of Ipatasertib on Day 1 and Day 8
Description: Plasma samples for pharmacokinetic characterization was collected at various timepoints in all participants.
Time Frame: 0.5 and 4 hours post dose on Day 1 of Cycle 1, 166 and 170 hours post dose from Day 1 of Cycle 1 (Cycle length = 28 days)
Population: The ITT population included all randomized participants. Reported here are data for participants with data available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ipatasertib + Paclitaxel
Number analyzed (Participants) | 73
ng/mL
  0.5 hours | 290 (312)
  4 hours: number analyzed (Participants) | 72
  4 hours | 196 (93.0)
  166 hours: number analyzed (Participants) | 71
  166 hours | 37.5 (28.3)
  170 hours: number analyzed (Participants) | 71
  170 hours | 355 (204)

14. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of Ipatasertib
Description: Plasma samples for pharmacokinetic characterization was collected on Day 1 and Day 8 in all participants.
Time Frame: as for outcome 13
Population: The ITT population included all participants.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ipatasertib + Paclitaxel
Number analyzed (Participants) | 76
ng/mL | 37.5 (28.3)

ADVERSE EVENTS:
Time Frame: 2 years and 6 months
Description: The safety population was identical to the ITT population. The ITT population comprised all 151 randomized patients.
Arm/Group | Ipatasertib + Paclitaxel | Placebo + Paclitaxel
All-Cause Mortality (participants affected / at risk) | 1/76 | 0/75
Serious Adverse Events (participants affected / at risk) | 10/76 | 3/75
Other Adverse Events (participants affected / at risk) | 76/76 | 73/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipatasertib + Paclitaxel (N=76) | Placebo + Paclitaxel (N=75)
Device related infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Complication associated with device (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipatasertib + Paclitaxel (N=76) | Placebo + Paclitaxel (N=75)
Anaemia (Blood and lymphatic system disorders) | 14 | 11
Neutropenia (Blood and lymphatic system disorders) | 7 | 6
Dry eye (Eye disorders) | 3 | 4
Lacrimation increased (Eye disorders) | 4 | 1
Abdominal distension (Gastrointestinal disorders) | 4 | 1
Abdominal Pain (Gastrointestinal disorders) | 14 | 6
Abdominal pain upper (Gastrointestinal disorders) | 7 | 4
Constipation (Gastrointestinal disorders) | 10 | 16
Diarrhoea (Gastrointestinal disorders) | 66 | 24
Dry mouth (Gastrointestinal disorders) | 7 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 8
Dyspepsia (Gastrointestinal disorders) | 12 | 9
Nausea (Gastrointestinal disorders) | 36 | 23
Stomatitis (Gastrointestinal disorders) | 5 | 6
Vomiting (Gastrointestinal disorders) | 17 | 4
Asthenia (General disorders) | 32 | 29
Fatigue (General disorders) | 23 | 24
Mucosal dryness (General disorders) | 4 | 0
Mucosal inflammation (General disorders) | 14 | 5
Oedema peripheral (General disorders) | 3 | 5
Pyrexia (General disorders) | 8 | 4
Conjunctivitis (Infections and infestations) | 2 | 5
Folliculitis (Infections and infestations) | 5 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 5
Urinary tract infection (Infections and infestations) | 8 | 9
Viral upper respiratory tract infection (Infections and infestations) | 4 | 7
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 4
Alanine aminotransferase increased (Investigations) | 5 | 5
Aspartate aminotransferase increased (Investigations) | 3 | 4
Neutrophil count decreased (Investigations) | 4 | 4
Decreased appetite (Metabolism and nutrition disorders) | 11 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 7
Dizziness (Nervous system disorders) | 7 | 8
Dysgeusia (Nervous system disorders) | 18 | 17
Hypoaesthesia (Nervous system disorders) | 1 | 4
Neuropathy peripheral (Nervous system disorders) | 14 | 14
Neurotoxicity (Nervous system disorders) | 9 | 6
Paraesthesia (Nervous system disorders) | 12 | 9
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 13
Anxiety (Psychiatric disorders) | 3 | 6
Insomnia (Psychiatric disorders) | 15 | 15
Dysuria (Renal and urinary disorders) | 1 | 5
Amenorrhoea (Reproductive system and breast disorders) | 1 | 5
Breast pain (Reproductive system and breast disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 40 | 40
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 4 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 3
Erythema (Skin and subcutaneous tissue disorders) | 5 | 4
Onycholysis (Skin and subcutaneous tissue disorders) | 5 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 10
Rash (Skin and subcutaneous tissue disorders) | 19 | 14
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 7
Flushing (Vascular disorders) | 7 | 4
Hot flush (Vascular disorders) | 6 | 5
Headache (Nervous system disorders) | 14 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT02301988/Prot_SAP_000.pdf